CLINICAL TRIAL: NCT01723839
Title: Phase II Clinical Protocol for the Treatment of Patients With Previously Untreated CLL With Four or Six Cycles of Fludarabine and Cyclophosphamide With Rituximab (FCR) Plus Lenalidomide Followed by Lenalidomide Consolidation/ Maintenance
Brief Title: Phase II Protocol for CLL With Fludarabine and Cyclophosphamide With Rituximab (FCR) Plus Lenalidomide
Acronym: FCR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hackensack Meridian Health (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00002262 RV-CLL-PI-0530
Record Dates: First submitted 2012-11-06; First posted 2012-11-08 (Estimated); Results first posted 2022-10-10 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Chronic Lymphocytic Leukemia (CLL)
Keywords: CLL; FCR; Rituximab; Lenalidomide; Cyclophosphamide
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — fludarabine; Cyclophosphamide; Rituximab; Lenalidomide; Receptors, Fc

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FCR with Lenalidomide (Other): Fludarabine, Cyclophosphamide, Rituximab, Lenalidomide - 19 subjects are treated in stage-1 with FCR plus 5mg lenalidomide increasing to 10mg and 15mg in subsequent cycles depending on toxicity. If there are at least 5 CRs after 4 cycles of FCR plus lenalidomide the study will accrue an additional 35 subjects.
  Interventions: Drug: Fludarabine, Cyclophosphamide, Rituximab, Lenalidomide

INTERVENTIONS:
Drug: Fludarabine, Cyclophosphamide, Rituximab, Lenalidomide — 19 subjects are treated in stage-1 with FCR plus 5mg lenalidomide increasing to 10mg and 15mg in subsequent cycles depending on toxicity.
  Other Names: FCR + Lenalidomide

SUMMARY:
In previously-untreated subjects with CLL, fludarabine and rituximab with or without cyclophosphamide (FR or FCR) produces complete responses (CR) of 40-80%. The major complication of FCR has been grade 3/4 neutropenia which was reduced using a lower dose of fludarabine and cyclophosphamide (FCR-Lite) The objective of this study is to evaluate the minimal residual disease (MRD) complete response rate (using the 2008 IWCLL guidelines) after 4 cycles of FCR-Lite plus lenalidomide in subjects with previously untreated CLL. Lenalidomide is active in frontline treatment of CLL as well as in patients with refractory disease. MRD has been demonstrated to be a sensitive surrogate marker for progression-free survival. If patients are MRD negative complete responders (CR) they will stop at 4 cycles of FCR-Lite followed by the lenalidomide consolidation/maintenance arm of the study. If they have a MRD positive CR or partial response (PR) they will continue with 2 additional cycles of FCR-Lite plus lenalidomide followed by lenalidomide consolidation/maintenance. They will be re-tested for MRD after the 6th cycle of FCR-Lite and after 6 and 12 months of lenalidomide monotherapy If they have no response (NR) or progressive disease (PD) following 4 cycles of FCR-Lite plus lenalidomide they will be removed from the study.

DETAILED DESCRIPTION:
STUDY OBJECTIVES:

Primary:

The primary objective is to evaluate the complete response rate following 4 cycles of FCR-Lite plus lenalidomide in previously untreated patients with CLL.

Secondary:

The first secondary objective is to evaluate the toxicity of patients with previously untreated CLL treated with FCR-Lite plus lenalidomide, followed by lenalidomide. The second is to evaluate the overall response rate and overall survival of patients with previously untreated CLL treated with FCR-Lite plus lenalidomide followed by lenalidomide. The third is to determine whether adding lenalidomide as a consolidation/maintenance therapy will eliminate bone marrow minimal residual disease in CR patients and whether patients who have a PR after 6 cycles of FCR-Lite plus lenalidomide will respond to 12 months of lenalidomide. The final secondary objective is to determine whether the expression of ZAP-70, CD38, and chromosomes correlate with response rate, duration of response, and survival for previously untreated patients with CLL.

STUDY DESIGN:

2-stage phase 2 study-design. 19 subjects are treated in stage-1 with FCR-Lite plus 5mg lenalidomide increasing to 10mg and 15mg in subsequent cycles depending on toxicity. If there are at least 5 CRs the study will accrue an additional 35 subjects (see statistical section). A secondary objective of this study will be to determine if MRD positive patients will become MRD negative with lenalidomide consolidation/maintenance and whether PR patients will convert to CRs Lenalidomide will begin 2 months after the last dose of FCR-Lite in all subjects with CR. It may begin as soon as 1 month after FCR-Lite plus lenalidomide in subjects with PR. Lenalidomide is given in 28 d cycles increasing the dose from 5 mg/d to 10 mg/d in cycle 2 and to 15mg in cycles 3-6 if well- tolerated (no grade-3 or -4 toxicity). Patients with creatinine clearance ≥30ml/min and <60ml/min will start at 2.5mg daily increasing to 5 and 10mg in subsequent cycles . Reduction to the prior dose is allowed for grade-3/-4 toxicity. MRD will be studied by flow cytometry from bone marrow and peripheral blood samples following 4 and 6 cycles of FCR-Lite and after 6 and 12 months of lenalidomide in CR patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have diagnosis of CLL (as defined by the NCI Criteria below:

  * Patients must have peripheral blood absolute lymphocyte count of >5,000/mm3 obtained within 2 weeks prior to start of study.
  * The lymphocytosis must consist of small, mature lymphocytes, with ≤55% (not greater than 55%) prolymphocytes.
* Patients must have phenotypically characterized CLL as defined as:

  1. The predominant population of cells share B-cell antigens with CD5 in the absence of other pan-T-cell markers (CD3, CD2, etc.);
  2. Surface immunoglobulin (slg) and CD20 with low-cell surface density expression.
  3. If surface immunoglobulin can be demonstrated, the leukemic cells are restricted to expression of either kappa or lambda.
* Splenomegaly, hepatomegaly or lymphadenopathy are not required for the diagnosis of CLL
* Patients must require chemotherapy
* Patients must not have received prior treatment cytotoxic, immunotherapy or investigational therapy.
* Patients must not have history of corticosteroid treatment for CLL, Autoimmune thrombocytopenia, or autoimmune hemolytic anemia.
* Calculated creatinine clearance ≥30ml/min by Cockcroft-Gault formula
* Bilirubin must be ≤1.5mg/dl, unless secondary to tumor, obtained within 2 weeks prior to registration
* Platelets ≥75x109/L, unless due to CLL involvement of bone marrow
* Neutrophils ≥1.5x109/L, unless due to CLL involvement of bone marrow
* AST or ALT < 2x upper limit of normal, unless related to CLL
* Age ≥18 years
* ECOG performance status 0-2
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test
* Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy
* Able to take aspirin (81mg or 325mg) daily as prophylactic anticoagulation
* Subject must provide written informed consent
* All study participants must be registered into the mandatory RevAssist® program, and be willing and able to comply with the requirements of RevAssist®

Exclusion Criteria:

* Patients with autoimmune hemolytic anemia or autoimmune thrombocytopenia are not eligible
* No prior immunotherapy, investigational or cytotoxic chemotherapy
* Patients with a history of steroid treatment for CLL/SLL autoimmune hemolytic anemia, or autoimmune thrombocytopenia are not eligible
* Patients with active infections requiring oral or intravenous (IV) antibiotics until resolution of the infection and completion of therapeutic antibiotics
* Women of childbearing potential and sexually active males who both refuse to use an accepted and effective method of contraception or women who are breastfeeding
* Patients with a second malignancy other than basal cell carcinoma or squamous cell carcinoma of the skin or in situ carcinoma of the cervix are not eligible unless the tumor was treated with curative intent at least two years previously
* History of known HIV
* History or presence CNS disease
* Evidence of laboratory TLS by Cairo-Bishop definition of Tumor Lysis Syndrome
* History of corticosteroid treatment for CLL, Autoimmune thrombocytopenia, or autoimmune hemolytic anemia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2012-02-22 (Actual); Primary Completion 2021-06-08 (Actual); Study Completion 2021-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andre Goy, MD, Principal Investigator — John Theurer Cancer Center at HackensackUMC
Locations (1):
- John Theurer Cancer Center at HackensackUMC, Hackensack, New Jersey, United States

REFERENCES:
- [Background] Rai KR, Patel DV. Chronic Lymphocytic Leukemia, in Hoffman R, Benz E, Shattil 5, Furie B, Cohen H, Silberstein L (eds): Hematology: Basic Principles and Practice, New York, Churchill Livingstone, 1995, p. 1308.
- [Background] Linet MS, Cartwright RA. Chronic lymphocytic leukemia: epidemiology and etiologic findings. Nouv Rev Fr Hematol (1978). 1988;30(5-6):353-7. PMID 3222144
- [Background] Jaksic B, Vitale B, Hauptmann E, Planinc-Peraica A, Ostojic S, Kusec R. The roles of age and sex in the prognosis of chronic leukaemias. A study of 373 cases. Br J Cancer. 1991 Aug;64(2):345-8. doi: 10.1038/bjc.1991.303. PMID 1892761
- [Background] Hallek M, Cheson BD, Catovsky D, Caligaris-Cappio F, Dighiero G, Dohner H, Hillmen P, Keating MJ, Montserrat E, Rai KR, Kipps TJ; International Workshop on Chronic Lymphocytic Leukemia. Guidelines for the diagnosis and treatment of chronic lymphocytic leukemia: a report from the International Workshop on Chronic Lymphocytic Leukemia updating the National Cancer Institute-Working Group 1996 guidelines. Blood. 2008 Jun 15;111(12):5446-56. doi: 10.1182/blood-2007-06-093906. Epub 2008 Jan 23. PMID 18216293
- [Background] Rai KR, Sawitsky A, Cronkite EP, Chanana AD, Levy RN, Pasternack BS. Clinical staging of chronic lymphocytic leukemia. Blood. 1975 Aug;46(2):219-34. PMID 1139039
- [Background] Rai KR, Sawitsky A. A review of the prognostic role of cytogenetic, phenotypic, morphologic, and immune function characteristics in chronic lymphocytic leukemia. Blood Cells. 1987;12(2):327-38. PMID 3304471
- [Background] Montserrat E, Rozman C. Bone marrow biopsy in chronic lymphocytic leukemia: a review of its prognostic importance. Blood Cells. 1987;12(2):315-26. PMID 3304470
- [Background] Montserrat E, Rozman C. Chronic lymphocytic leukaemia: prognostic factors and natural history. Baillieres Clin Haematol. 1993 Dec;6(4):849-66. doi: 10.1016/s0950-3536(05)80179-9. PMID 8038493
- [Background] Han T, Bhargava A, Henderson ES, et al. Prognostic significance of beta-2-microglobulin (-2m) in chronic lymphocytic leukemia (CLL) and non-Hodgkin's lymphoma (NHL). Proc Amer Soc Clin Oncol 1989; 8:270 (abstr 270).
- [Background] Montserrat E, Alcala A, Parody R, Domingo A, Garcia-Conde J, Bueno J, Ferran C, Sanz MA, Giralt M, Rubio D, et al. Treatment of chronic lymphocytic leukemia in advanced stages. A randomized trial comparing chlorambucil plus prednisone versus cyclophosphamide, vincristine, and prednisone. Cancer. 1985 Nov 15;56(10):2369-75. doi: 10.1002/1097-0142(19851115)56:103.0.co;2-n. PMID 3899346
- [Background] Fais F, Ghiotto F, Hashimoto S, Sellars B, Valetto A, Allen SL, Schulman P, Vinciguerra VP, Rai K, Rassenti LZ, Kipps TJ, Dighiero G, Schroeder HW Jr, Ferrarini M, Chiorazzi N. Chronic lymphocytic leukemia B cells express restricted sets of mutated and unmutated antigen receptors. J Clin Invest. 1998 Oct 15;102(8):1515-25. doi: 10.1172/JCI3009. PMID 9788964
- [Background] Damle RN, Wasil T, Fais F, Ghiotto F, Valetto A, Allen SL, Buchbinder A, Budman D, Dittmar K, Kolitz J, Lichtman SM, Schulman P, Vinciguerra VP, Rai KR, Ferrarini M, Chiorazzi N. Ig V gene mutation status and CD38 expression as novel prognostic indicators in chronic lymphocytic leukemia. Blood. 1999 Sep 15;94(6):1840-7. PMID 10477712
- [Background] Oscier DG, Thompsett A, Zhu D, Stevenson FK. Differential rates of somatic hypermutation in V(H) genes among subsets of chronic lymphocytic leukemia defined by chromosomal abnormalities. Blood. 1997 Jun 1;89(11):4153-60. PMID 9166858
- [Background] Hamblin TJ, Davis Z, Gardiner A, Oscier DG, Stevenson FK. Unmutated Ig V(H) genes are associated with a more aggressive form of chronic lymphocytic leukemia. Blood. 1999 Sep 15;94(6):1848-54. PMID 10477713
- [Background] Crespo M, Bosch F, Villamor N, Bellosillo B, Colomer D, Rozman M, Marce S, Lopez-Guillermo A, Campo E, Montserrat E. ZAP-70 expression as a surrogate for immunoglobulin-variable-region mutations in chronic lymphocytic leukemia. N Engl J Med. 2003 May 1;348(18):1764-75. doi: 10.1056/NEJMoa023143. PMID 12724482
- [Background] Lin K, Sherrington PD, Dennis M, Matrai Z, Cawley JC, Pettitt AR. Relationship between p53 dysfunction, CD38 expression, and IgV(H) mutation in chronic lymphocytic leukemia. Blood. 2002 Aug 15;100(4):1404-9. doi: 10.1182/blood-2001-11-0066. PMID 12149224
- [Background] Gahrton G, Juliusson G. Clinical implication of chromosomal aberrations in chronic B-lymphocytic leukaemia cells. Nouv Rev Fr Hematol (1978). 1988;30(5-6):389-92. PMID 3265508
- [Background] Bird ML, Ueshima Y, Rowley JD, Haren JM, Vardiman JW. Chromosome abnormalities in B cell chronic lymphocytic leukemia and their clinical correlations. Leukemia. 1989 Mar;3(3):182-91. PMID 2918755
- [Background] Krober A, Seiler T, Benner A, Bullinger L, Bruckle E, Lichter P, Dohner H, Stilgenbauer S. V(H) mutation status, CD38 expression level, genomic aberrations, and survival in chronic lymphocytic leukemia. Blood. 2002 Aug 15;100(4):1410-6. PMID 12149225
- [Background] Rozman C, Montserrat E. Bone marrow biopsy in chronic lymphocytic leukemia. Nouv Rev Fr Hematol (1978). 1988;30(5-6):369-71. PMID 3065734
- [Background] Pangalis GA, Boussiotis VA, Kittas C. B-chronic lymphocytic leukemia. Disease progression in 150 untreated stage A and B patients as predicted by bone marrow pattern. Nouv Rev Fr Hematol (1978). 1988;30(5-6):373-5. PMID 3222147
- [Background] Montserrat E, Vinolas N, Reverter JC, Rozman C. Natural history of chronic lymphocytic leukemia: on the progression and progression and prognosis of early clinical stages. Nouv Rev Fr Hematol (1978). 1988;30(5-6):359-61. PMID 3222145
- [Background] Shustik C, Mick R, Silver R, Sawitsky A, Rai K, Shapiro L. Treatment of early chronic lymphocytic leukemia: intermittent chlorambucil versus observation. Hematol Oncol. 1988 Jan-Mar;6(1):7-12. doi: 10.1002/hon.2900060103. PMID 3277904
- [Background] Liepman M, Votaw ML. The treatment of chronic lymphocytic leukemia with COP chemotherapy. Cancer. 1978 May;41(5):1664-9. doi: 10.1002/1097-0142(197805)41:53.0.co;2-q. PMID 647620
- [Background] Oken MM, Kaplan ME. Combination chemotherapy with cyclophosphamide, vincristine, and prednisone in the treatment of refractory chronic lymphocytic leukemia. Cancer Treat Rep. 1979 Mar;63(3):441-7. No abstract available. PMID 371799
- [Background] Hansen MM, Andersen E, Christensen BE, Christiansen I, Geisler C, Kristensen D, Jensen KB, Junker P. CHOP versus prednisolone + chlorambucil in chronic lymphocytic leukemia (CLL): preliminary results of a randomized multicenter study. Nouv Rev Fr Hematol (1978). 1988;30(5-6):433-6. PMID 3065739
- [Background] Raphael B, Andersen JW, Silber R, Oken M, Moore D, Bennett J, Bonner H, Hahn R, Knospe WH, Mazza J, et al. Comparison of chlorambucil and prednisone versus cyclophosphamide, vincristine, and prednisone as initial treatment for chronic lymphocytic leukemia: long-term follow-up of an Eastern Cooperative Oncology Group randomized clinical trial. J Clin Oncol. 1991 May;9(5):770-6. doi: 10.1200/JCO.1991.9.5.770. PMID 2016618
- [Background] Grever MR, Kopecky KJ, Coltman CA, Files JC, Greenberg BR, Hutton JJ, Talley R, Von Hoff DD, Balcerzak SP. Fludarabine monophosphate: a potentially useful agent in chronic lymphocytic leukemia. Nouv Rev Fr Hematol (1978). 1988;30(5-6):457-9. PMID 2464793
- [Background] Keating MJ, Kantarjian H, O'Brien S, Koller C, Talpaz M, Schachner J, Childs CC, Freireich EJ, McCredie KB. Fludarabine: a new agent with marked cytoreductive activity in untreated chronic lymphocytic leukemia. J Clin Oncol. 1991 Jan;9(1):44-9. doi: 10.1200/JCO.1991.9.1.44. PMID 1702145
- [Background] Rai KR, Peterson BL, Appelbaum FR, Kolitz J, Elias L, Shepherd L, Hines J, Threatte GA, Larson RA, Cheson BD, Schiffer CA. Fludarabine compared with chlorambucil as primary therapy for chronic lymphocytic leukemia. N Engl J Med. 2000 Dec 14;343(24):1750-7. doi: 10.1056/NEJM200012143432402. PMID 11114313
- [Background] O'Brien S, Kantarjian H, Beran M, Smith T, Koller C, Estey E, Robertson LE, Lerner S, Keating M. Results of fludarabine and prednisone therapy in 264 patients with chronic lymphocytic leukemia with multivariate analysis-derived prognostic model for response to treatment. Blood. 1993 Sep 15;82(6):1695-700. PMID 8400226
- [Background] Anaissie E, Kontoyiannis DP, Kantarjian H, Elting L, Robertson LE, Keating M. Listeriosis in patients with chronic lymphocytic leukemia who were treated with fludarabine and prednisone. Ann Intern Med. 1992 Sep 15;117(6):466-9. doi: 10.7326/0003-4819-117-6-466. PMID 1354425
- [Background] Johnston JB, Verburg L, Shore T, Williams M, Israels LG, Begleiter A. Combination therapy with nucleoside analogs and alkylating agents. Leukemia. 1994 Apr;8 Suppl 1:S140-3. PMID 8152282
- [Background] Begleiter A, Pugh L, Israels LG, Johnston JB. Enhanced cytotoxicity and inhibition of DNA damage repair in irradiated murine L5178Y lymphoblasts and human chronic lymphocytic leukemia cells treated with 2'-deoxycoformycin and deoxyadenosine in vitro. Cancer Res. 1988 Jul 15;48(14):3981-6. PMID 3260129
- [Background] O'Brien SM, Kantarjian HM, Cortes J, Beran M, Koller CA, Giles FJ, Lerner S, Keating M. Results of the fludarabine and cyclophosphamide combination regimen in chronic lymphocytic leukemia. J Clin Oncol. 2001 Mar 1;19(5):1414-20. doi: 10.1200/JCO.2001.19.5.1414. PMID 11230486
- [Background] Flinn IW, Byrd JC, Morrison C, Jamison J, Diehl LF, Murphy T, Piantadosi S, Seifter E, Ambinder RF, Vogelsang G, Grever MR. Fludarabine and cyclophosphamide with filgrastim support in patients with previously untreated indolent lymphoid malignancies. Blood. 2000 Jul 1;96(1):71-5. PMID 10891432
- [Background] Hainsworth JD, Litchy S, Barton JH, Houston GA, Hermann RC, Bradof JE, Greco FA; Minnie Pearl Cancer Research Network. Single-agent rituximab as first-line and maintenance treatment for patients with chronic lymphocytic leukemia or small lymphocytic lymphoma: a phase II trial of the Minnie Pearl Cancer Research Network. J Clin Oncol. 2003 May 1;21(9):1746-51. doi: 10.1200/JCO.2003.09.027. PMID 12721250
- [Background] O'Brien SM, Kantarjian H, Thomas DA, Giles FJ, Freireich EJ, Cortes J, Lerner S, Keating MJ. Rituximab dose-escalation trial in chronic lymphocytic leukemia. J Clin Oncol. 2001 Apr 15;19(8):2165-70. doi: 10.1200/JCO.2001.19.8.2165. PMID 11304768
- [Background] Byrd JC, Murphy T, Howard RS, Lucas MS, Goodrich A, Park K, Pearson M, Waselenko JK, Ling G, Grever MR, Grillo-Lopez AJ, Rosenberg J, Kunkel L, Flinn IW. Rituximab using a thrice weekly dosing schedule in B-cell chronic lymphocytic leukemia and small lymphocytic lymphoma demonstrates clinical activity and acceptable toxicity. J Clin Oncol. 2001 Apr 15;19(8):2153-64. doi: 10.1200/JCO.2001.19.8.2153. PMID 11304767
- [Background] Ladetto M, Bergui L, Ricca I, Campana S, Pileri A, Tarella C. Rituximab anti-CD20 monoclonal antibody induces marked but transient reductions of peripheral blood lymphocytes in chronic lymphocytic leukaemia patients. Med Oncol. 2000 Aug;17(3):203-10. doi: 10.1007/BF02780529. PMID 10962531
- [Background] Huhn D, von Schilling C, Wilhelm M, Ho AD, Hallek M, Kuse R, Knauf W, Riedel U, Hinke A, Srock S, Serke S, Peschel C, Emmerich B; German Chronic Lymphocytic Leukemia Study Group. Rituximab therapy of patients with B-cell chronic lymphocytic leukemia. Blood. 2001 Sep 1;98(5):1326-31. doi: 10.1182/blood.v98.5.1326. PMID 11520778
- [Background] List A, Kurtin S, Roe DJ, Buresh A, Mahadevan D, Fuchs D, Rimsza L, Heaton R, Knight R, Zeldis JB. Efficacy of lenalidomide in myelodysplastic syndromes. N Engl J Med. 2005 Feb 10;352(6):549-57. doi: 10.1056/NEJMoa041668. PMID 15703420
- [Background] List A, Dewald G, Bennett J, Giagounidis A, Raza A, Feldman E, Powell B, Greenberg P, Thomas D, Stone R, Reeder C, Wride K, Patin J, Schmidt M, Zeldis J, Knight R; Myelodysplastic Syndrome-003 Study Investigators. Lenalidomide in the myelodysplastic syndrome with chromosome 5q deletion. N Engl J Med. 2006 Oct 5;355(14):1456-65. doi: 10.1056/NEJMoa061292. PMID 17021321
- [Background] Richardson PG, Schlossman RL, Weller E, Hideshima T, Mitsiades C, Davies F, LeBlanc R, Catley LP, Doss D, Kelly K, McKenney M, Mechlowicz J, Freeman A, Deocampo R, Rich R, Ryoo JJ, Chauhan D, Balinski K, Zeldis J, Anderson KC. Immunomodulatory drug CC-5013 overcomes drug resistance and is well tolerated in patients with relapsed multiple myeloma. Blood. 2002 Nov 1;100(9):3063-7. doi: 10.1182/blood-2002-03-0996. PMID 12384400
- [Background] Richardson PG, Blood E, Mitsiades CS, Jagannath S, Zeldenrust SR, Alsina M, Schlossman RL, Rajkumar SV, Desikan KR, Hideshima T, Munshi NC, Kelly-Colson K, Doss D, McKenney ML, Gorelik S, Warren D, Freeman A, Rich R, Wu A, Olesnyckyj M, Wride K, Dalton WS, Zeldis J, Knight R, Weller E, Anderson KC. A randomized phase 2 study of lenalidomide therapy for patients with relapsed or relapsed and refractory multiple myeloma. Blood. 2006 Nov 15;108(10):3458-64. doi: 10.1182/blood-2006-04-015909. Epub 2006 Jul 13. PMID 16840727
- [Background] Rajkumar SV, Hayman SR, Lacy MQ, Dispenzieri A, Geyer SM, Kabat B, Zeldenrust SR, Kumar S, Greipp PR, Fonseca R, Lust JA, Russell SJ, Kyle RA, Witzig TE, Gertz MA. Combination therapy with lenalidomide plus dexamethasone (Rev/Dex) for newly diagnosed myeloma. Blood. 2005 Dec 15;106(13):4050-3. doi: 10.1182/blood-2005-07-2817. Epub 2005 Aug 23. PMID 16118317
- [Background] Marriott JB, Clarke IA, Dredge K, Muller G, Stirling D, Dalgleish AG. Thalidomide and its analogues have distinct and opposing effects on TNF-alpha and TNFR2 during co-stimulation of both CD4(+) and CD8(+) T cells. Clin Exp Immunol. 2002 Oct;130(1):75-84. doi: 10.1046/j.1365-2249.2002.01954.x. PMID 12296856
- [Background] Mangiameli DP, Blansfield JA, Kachala S, Lorang D, Schafer PH, Muller GW, Stirling DI, Libutti SK. Combination therapy targeting the tumor microenvironment is effective in a model of human ocular melanoma. J Transl Med. 2007 Jul 18;5:38. doi: 10.1186/1479-5876-5-38. PMID 17640369
- [Background] Tai YT, Li XF, Catley L, Coffey R, Breitkreutz I, Bae J, Song W, Podar K, Hideshima T, Chauhan D, Schlossman R, Richardson P, Treon SP, Grewal IS, Munshi NC, Anderson KC. Immunomodulatory drug lenalidomide (CC-5013, IMiD3) augments anti-CD40 SGN-40-induced cytotoxicity in human multiple myeloma: clinical implications. Cancer Res. 2005 Dec 15;65(24):11712-20. doi: 10.1158/0008-5472.CAN-05-1657. PMID 16357183
- [Background] LeBlanc R, Hideshima T, Catley LP, Shringarpure R, Burger R, Mitsiades N, Mitsiades C, Cheema P, Chauhan D, Richardson PG, Anderson KC, Munshi NC. Immunomodulatory drug costimulates T cells via the B7-CD28 pathway. Blood. 2004 Mar 1;103(5):1787-90. doi: 10.1182/blood-2003-02-0361. Epub 2003 Sep 25. PMID 14512311
- [Background] Hernandez-Ilizaliturri FJ, Reddy N, Holkova B, Ottman E, Czuczman MS. Immunomodulatory drug CC-5013 or CC-4047 and rituximab enhance antitumor activity in a severe combined immunodeficient mouse lymphoma model. Clin Cancer Res. 2005 Aug 15;11(16):5984-92. doi: 10.1158/1078-0432.CCR-05-0577. PMID 16115943
- [Background] Pellagatti A, Jadersten M, Forsblom AM, Cattan H, Christensson B, Emanuelsson EK, Merup M, Nilsson L, Samuelsson J, Sander B, Wainscoat JS, Boultwood J, Hellstrom-Lindberg E. Lenalidomide inhibits the malignant clone and up-regulates the SPARC gene mapping to the commonly deleted region in 5q- syndrome patients. Proc Natl Acad Sci U S A. 2007 Jul 3;104(27):11406-11. doi: 10.1073/pnas.0610477104. Epub 2007 Jun 18. PMID 17576924
- [Background] Chanan-Khan A, Miller KC, Musial L, Lawrence D, Padmanabhan S, Takeshita K, Porter CW, Goodrich DW, Bernstein ZP, Wallace P, Spaner D, Mohr A, Byrne C, Hernandez-Ilizaliturri F, Chrystal C, Starostik P, Czuczman MS. Clinical efficacy of lenalidomide in patients with relapsed or refractory chronic lymphocytic leukemia: results of a phase II study. J Clin Oncol. 2006 Dec 1;24(34):5343-9. doi: 10.1200/JCO.2005.05.0401. Epub 2006 Nov 6. PMID 17088571
- [Background] Ferrajoli A, Lee BN, Schlette EJ, O'Brien SM, Gao H, Wen S, Wierda WG, Estrov Z, Faderl S, Cohen EN, Li C, Reuben JM, Keating MJ. Lenalidomide induces complete and partial remissions in patients with relapsed and refractory chronic lymphocytic leukemia. Blood. 2008 Jun 1;111(11):5291-7. doi: 10.1182/blood-2007-12-130120. Epub 2008 Mar 11. PMID 18334676
- [Background] Andritsos LA, Johnson AJ, Lozanski G, Blum W, Kefauver C, Awan F, Smith LL, Lapalombella R, May SE, Raymond CA, Wang DS, Knight RD, Ruppert AS, Lehman A, Jarjoura D, Chen CS, Byrd JC. Higher doses of lenalidomide are associated with unacceptable toxicity including life-threatening tumor flare in patients with chronic lymphocytic leukemia. J Clin Oncol. 2008 May 20;26(15):2519-25. doi: 10.1200/JCO.2007.13.9709. Epub 2008 Apr 21. PMID 18427150
- [Background] Chen C, Paul H, Xu W, et al: A phase II study of lenalidomide in previously untreated, symptomatic chronic lymphocytic leukemia (CLL). Blood 112:23, 2008 (abstr 44).
- [Background] Byrd JC, Peterson BL, Morrison VA, Park K, Jacobson R, Hoke E, Vardiman JW, Rai K, Schiffer CA, Larson RA. Randomized phase 2 study of fludarabine with concurrent versus sequential treatment with rituximab in symptomatic, untreated patients with B-cell chronic lymphocytic leukemia: results from Cancer and Leukemia Group B 9712 (CALGB 9712). Blood. 2003 Jan 1;101(1):6-14. doi: 10.1182/blood-2002-04-1258. Epub 2002 Jul 5. PMID 12393429
- [Background] Hallek M, Fischer K, Fingerle-Rowson G, Fink AM, Busch R, Mayer J, Hensel M, Hopfinger G, Hess G, von Grunhagen U, Bergmann M, Catalano J, Zinzani PL, Caligaris-Cappio F, Seymour JF, Berrebi A, Jager U, Cazin B, Trneny M, Westermann A, Wendtner CM, Eichhorst BF, Staib P, Buhler A, Winkler D, Zenz T, Bottcher S, Ritgen M, Mendila M, Kneba M, Dohner H, Stilgenbauer S; International Group of Investigators; German Chronic Lymphocytic Leukaemia Study Group. Addition of rituximab to fludarabine and cyclophosphamide in patients with chronic lymphocytic leukaemia: a randomised, open-label, phase 3 trial. Lancet. 2010 Oct 2;376(9747):1164-74. doi: 10.1016/S0140-6736(10)61381-5. PMID 20888994
- [Background] Keating MJ, O'Brien S, Albitar M, Lerner S, Plunkett W, Giles F, Andreeff M, Cortes J, Faderl S, Thomas D, Koller C, Wierda W, Detry MA, Lynn A, Kantarjian H. Early results of a chemoimmunotherapy regimen of fludarabine, cyclophosphamide, and rituximab as initial therapy for chronic lymphocytic leukemia. J Clin Oncol. 2005 Jun 20;23(18):4079-88. doi: 10.1200/JCO.2005.12.051. Epub 2005 Mar 14. PMID 15767648
- [Background] Brown JR, Abramson J, Hochberg E, Mikler E, Dalton V, Werner L, Reynolds H, Thompson C, McDonough SM, Kuang Y, Ritz J, Neuberg D, Freedman AS. A phase I study of lenalidomide in combination with fludarabine and rituximab in previously untreated CLL/SLL. Leukemia. 2010 Nov;24(11):1972-5. doi: 10.1038/leu.2010.199. Epub 2010 Sep 16. No abstract available. PMID 20844565
- [Background] Provan D, Bartlett-Pandite L, Zwicky C, Neuberg D, Maddocks A, Corradini P, Soiffer R, Ritz J, Nadler LM, Gribben JG. Eradication of polymerase chain reaction-detectable chronic lymphocytic leukemia cells is associated with improved outcome after bone marrow transplantation. Blood. 1996 Sep 15;88(6):2228-35. PMID 8822943
- [Background] Moreton P, Kennedy B, Lucas G, Leach M, Rassam SM, Haynes A, Tighe J, Oscier D, Fegan C, Rawstron A, Hillmen P. Eradication of minimal residual disease in B-cell chronic lymphocytic leukemia after alemtuzumab therapy is associated with prolonged survival. J Clin Oncol. 2005 May 1;23(13):2971-9. doi: 10.1200/JCO.2005.04.021. Epub 2005 Feb 28. PMID 15738539
- [Background] Bosch F, Ferrer A, Lopez-Guillermo A, Gine E, Bellosillo B, Villamor N, Colomer D, Cobo F, Perales M, Esteve J, Altes A, Besalduch J, Ribera JM, Montserrat E; GELCAB (Grup per l'Estudi dels Limfomes a Catalunya i Balears). Fludarabine, cyclophosphamide and mitoxantrone in the treatment of resistant or relapsed chronic lymphocytic leukaemia. Br J Haematol. 2002 Dec;119(4):976-84. doi: 10.1046/j.1365-2141.2002.03959.x. PMID 12472576
- [Background] Boettcher S, Fischer K, Stilgenbauer S, Busch R, Fingerle-Rowson G, Fink AM et al. Quantitative MRD assessments predict progression-free survival in CLL patients treated with fludarabine and cyclophosphamide with or without rituximab - a prospective analysis in 471 patients from the randomized GCLLSG CLL8 trial. Blood 2008; 112: 11, abstract 326)
- [Background] Kay NE, Geyer SM, Call TG, Shanafelt TD, Zent CS, Jelinek DF, Tschumper R, Bone ND, Dewald GW, Lin TS, Heerema NA, Smith L, Grever MR, Byrd JC. Combination chemoimmunotherapy with pentostatin, cyclophosphamide, and rituximab shows significant clinical activity with low accompanying toxicity in previously untreated B chronic lymphocytic leukemia. Blood. 2007 Jan 15;109(2):405-11. doi: 10.1182/blood-2006-07-033274. Epub 2006 Sep 28. PMID 17008537
- [Background] Foon KA, Boyiadzis M, Land SR, Marks S, Raptis A, Pietragallo L, Meisner D, Laman A, Sulecki M, Butchko A, Schaefer P, Lenzer D, Tarhini A. Chemoimmunotherapy with low-dose fludarabine and cyclophosphamide and high dose rituximab in previously untreated patients with chronic lymphocytic leukemia. J Clin Oncol. 2009 Feb 1;27(4):498-503. doi: 10.1200/JCO.2008.17.2619. Epub 2008 Dec 15. PMID 19075274
- [Background] Simon R. Optimal two-stage designs for phase II clinical trials. Control Clin Trials. 1989 Mar;10(1):1-10. doi: 10.1016/0197-2456(89)90015-9. PMID 2702835
- [Background] Dufy DE, Santner TJ, Confidence intervals for binomial parameter based on multistage tests. Biometrics 43:81-93, 1987.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | FCR With Lenalidomide
Started | 21
Completed | 12
Not Completed | 9

BASELINE CHARACTERISTICS:
Arm/Group | FCR With Lenalidomide
Number analyzed (Participants) | 21
Age, Continuous [Median (Full Range); unit: years] | 62.5 [42 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 18
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Complete Response
Description: Analysis of the Primary Endpoint: The complete responses will be estimated by the number of patients with CR divided by the total number of evaluable patients.
Time Frame: 28 day cycle, up to 4 cycles
Population: Of the 21 were enrolled, 20 were eligible for response evaluation.
Measure: Number; unit: Percentage of Participants
Arm/Group | FCR With Lenalidomide
Number analyzed (Participants) | 20
Percentage of Participants | 45

2. Secondary Outcome: Overall Response Rate
Description: Analysis of the other Secondary Endpoints: The overall response rate will be estimated by the number of patients with complete and partial responses divided by the total number of evaluable patients.
Time Frame: 28 day cycle, up to 6 cycles
Population: Of the 21 were enrolled, 20 were eligible for response evaluation.
Measure: Number; unit: Percentage of Participants
Arm/Group | FCR With Lenalidomide
Number analyzed (Participants) | 20
Percentage of Participants | 95

ADVERSE EVENTS:
Time Frame: From study enrollment to end of treatment, up to 18 months
Arm/Group | FCR With Lenalidomide
All-Cause Mortality (participants affected / at risk) | 1/21
Serious Adverse Events (participants affected / at risk) | 9/21
Other Adverse Events (participants affected / at risk) | 19/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FCR With Lenalidomide (N=21)
Maculopapular Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Neutropenic Fever (Blood and lymphatic system disorders) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bilateral Leg Weakness (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FCR With Lenalidomide (N=21)
Leukopenia (Blood and lymphatic system disorders) | 13 (13)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 19 (33)
Hyperglycemia (Blood and lymphatic system disorders) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Infusion Reaction (Blood and lymphatic system disorders) | 1 (1)
Bacteremia (Infections and infestations) | 1 (1)
Pustular Rash (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-03-14): https://cdn.clinicaltrials.gov/large-docs/39/NCT01723839/Prot_SAP_000.pdf